CLINICAL TRIAL: NCT05454527
Title: Follow-up of a Cohort of Patients With Inflammatory Myopathies Associated With a Biobank: MASC 2 Project (Myositis, Muscles, DNA/RNA Serum Cells)
Brief Title: Follow-up of Patients With Inflammatory Myopathies Associated With a Biobank
Acronym: MASC2
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220491
Record Dates: First submitted 2022-06-17; First posted 2022-07-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Myositis; Idiopathic Inflammatory Myositis; Drug-induced Inflammatory Myositis
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — biopsy residual samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myositis are rare diseases for which the development of a cohort associated with a bank of biological samples (biobank) will allow for the conduct of researches to better delineate the underlying pathophysiology and find cures. This prospective cohort of patients with myositis will allow for identification of factors favouring the occurrence of myositis, whether they are constitutional (genetic) or acquired (environmental or drug). Different subgroups of myositis used for prognostication will be identified based on clinico-demographical variables, the nature of the organs involved beyond peripheral muscles (cardiac, diaphragm) and biomarkers abnormalities

DETAILED DESCRIPTION:
Myositis is a rare autoimmune disease in which the immune system mistakenly attacks the patient's own peripheral muscles. This aggression manifests by muscle inflammation and necrosis responsible for a motor deficit of varying severity. The treatments available today are insufficient and are non-specific. Biological criteria, issued from simple blood or muscle tests are missing, and they will help to define the activity of the disease and the efficacy of treatments. The MASC protocol will include patients with myositis, and investigators will collect clinical, radiological, electrophysiological, histological and biological data to be used for researches aiming at better understanding this entity. A biobank (muscle biopsy, DNA, serum, plasma, PBMCs) will be acquired on this prospective cohort. The study itself will be composed of a baseline visit and monthly to yearly follow-up visits which will assess:

* Clinical examination with an evaluation of the muscle strength and function impairment/handicap, including but not limited to:
* Manual testing of proximal axial and distal muscles on the five points Medical Research Council (MRC) scale
* Barré tests and Mingazzini tests, number of stand-up / sitting, leg crossing
* Biometry, lab and radiological measurements: muscle enzymes (creatine phosphokinase CPK, troponin, C-reactive protein, quantification of autoantibodies, muscle MRI, muscle biopsy, thorax tomodensitometry, pulmonary test function
* Extra-muscular evaluation: cardiac examination and work-up (echocardiography, cardiac MRI and Positron Emission Tomography (PET) scanner, cardiac biopsies), pulmonary evaluation, rheumatological and dermatological assessment, history of thromboembolic disease and cancer Patient activity assessment: evaluation of daily life activity by both patient and physician using a Visual Analogue Scale
* Quality of life questionnaires
* Evaluation of the efficacy and toxicity of specific treatments For each patient, the date of last visit or contact will be collected as well as outcomes, particularly for the cause of death if relevant. Data from the biobank MASC " Muscles DNA/RNA Serum and Cells " will be added to other data. The biobank has been fully registered with local authorities and ethical committees ("Committee for Personal Protection (CPP)" CPP agreement). It contains peripheral blood mononuclear cells (PBMC), serum, DNA and RNA from blood and muscular biopsies collected at the diagnosis stage. The database contains immunological and genetical data.

This prospective study will also aim at:

* Identify the differential pathophysiological processes between the different subgroups of myositis
* Identify prognostic factors, including the different treatment modalities used
* Improve physiopathological knowledge (clinico-anatomobiological characteristics and identification of other biomarkers through the biobank)
* Improve the evaluation of the clinical outcomes/endpoints for future trials
* Develop clinical trials for homogeneous subgroups of patients, based on their pathophysiology and evaluated on the appropriate endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suspicion of Myositis defined according to reference classifications: Dermatomyositis (DM), polymyositis (PM) defined as early as 1975 by Bohan and Peter, inclusion myositis (IM) according to the criteria of Griggs et al, 1995 and autoimmune necrotizing myopathy (ANM) by Hoogendijk et al, in 2004 and iatrogenic (e.g. drug-induced) myositis.
* No opposition from patients to the use of their data
* Signature of consents for the constitution of the biobank and the genetic analyses

Exclusion Criteria:

* Patients under AME
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with myositis included during consultation visits or routine hospitalizations in the Internal Medicine Department, Reference Center for Neuromuscular Pathology, at the Pitié Salpêtrière Hospital
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2057-10-26 (Estimated); Study Completion 2057-10-26 (Estimated)

PRIMARY OUTCOMES:
Characterisation of the different myositis subgroups based on clinical, radiological, electrophysiological and histobiological evaluations | baseline: first 30 days after inclusion
  Characterisation of the different myositis subgroups based on clinical, radiological, electrophysiological and histobiological evaluations

SECONDARY OUTCOMES:
Characterisation of the natural history of myositis subgroups :responses to treatments, prognosis factors, evolution | up to twenty years after inclusion
  Characterisation of the natural history of myositis subgroups :responses to treatments, prognosis factors, evolution
Characterisation of an immune system signature, using peripheral blood mononuclear cells and muscular biopsies, DNA and RNA sequencing, and autoantibodies | baseline: first 30 days after inclusion
  Characterisation of an immune system signature, using peripheral blood mononuclear cells and muscular biopsies, DNA and RNA sequencing, and autoantibodies
Risk factors for All-cause mortality depending on patient's and disease characteristics | up to twenty years after inclusion
  Risk factors for All-cause mortality depending on patient's and disease characteristics including clinical, radiological electrophysiological, histo-biological and immunological as well as treatment received stratified by each subgroup of myositis
Change of the quality of life, using quality of life questionnaires, depending of patients and disease characteristics | up to twenty years after inclusion
  Change of the quality of life, using quality of life questionnaires, depending of patients and disease characteristics (HAQ (Health Assessment Questionnaire)global health status scale (0-100))
Change of activity impairment using an evaluation of daily life activity by both patient and physician using a Visual Analogue Scale depending of patients and disease characteristics | up to twenty years after inclusion
  Using analogue Scale depending of patients and disease characteristics:
  Physician's assessment of disease activity in the muscle area (VAS 0-10) Physician's evaluation of the disease activity in the skin area (VAS 0-10) Physician's evaluation of general signs of disease activity (VAS 0-10) Physician's assessment of disease activity in rheumatology (VAS 0-10) Physician's assessment of disease activity in the digestive area (VAS 0-10) Physician's assessment of disease activity in the pulmonary area (VAS 0-10) Physician's assessment of disease activity in the cardiac area (VAS 0-10) Doctor's assessment of disease activity in the extra-muscular area (VAS 0-10) Overall evaluation of the disease activity (muscular and extra-muscular) by the PHYSICIAN (VAS 0-10) Global evaluation of the disease activity by the PATIENT (VAS 0-10)
Characterisation of a quality-of-life scale using biological data (CPK), muscle weakness (muscle testing) and other visceral involvements | up to twenty years after inclusion
  Using MM8 testing (0-150) visceral involvements
Characterisation of a global activity scale using biological data (CPK), muscle weakness (muscle testing) and other visceral involvements | up to twenty years after inclusion
  Using MM8 testing (0-150)
Incidence of major cardio-vascular events | up to twenty years after inclusion
  Incidence of major cardio-vascular events
Consequences on outcomes of major cardio-vascular events | up to twenty years after inclusion
  Major cardiovascular will include:
  * Heart failure
  * Myocardial infarction
  * Stroke
  * Sudden cardiac death
  * High-degree atrio-ventricular blocks
  * High-degree sinus dysfunction
  * Sustained ventricular tachycardia
Correlation of myositis with the development of extra-muscular diseases including but not limited to dermatological, rheumatological, cardiological and pneumological associated diseases | up to twenty years after inclusion
  Correlation of myositis with the development of extra-muscular diseases including but not limited to dermatological, rheumatological, cardiological and pneumological associated diseases
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using spirometry (Vital capacity in the sitting position)
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Vital capacity in supine position)
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (FEV1/VC ratio)
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Total lung capacity by Plethysmographic)
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Inspiratory capacity)
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (maximum static inspiratory pressure as % of predicted value)
Characterisation of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Sniff nasal inspiratory pressure in % of predicted value)
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Vital capacity in the sitting position )
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry ( Vital capacity in supine position )
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (FEV1/VC ratio)
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Total lung capacity by Plethysmographic)
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Inspiratory capacity)
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (maximum static inspiratory pressure as % of predicted value)
Characterisation of diaphragmatic failure with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Sniff nasal inspiratory pressure in % of predicted value)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Vital capacity in supine position)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Vital capacity in the sitting position)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (FEV1/VC ratio)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Total lung capacity by Plethysmographic)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Inspiratory capacity)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (maximum static inspiratory pressure as % of predicted value)
Follow up of respiratory function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Sniff nasal inspiratory pressure in % of predicted value)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Sniff nasal inspiratory pressure in % of predicted value)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (maximum static inspiratory pressure as % of predicted value)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Inspiratory capacity)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Total lung capacity by Plethysmographic)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (FEV1/VC ratio)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Vital capacity in the sitting position)
Follow up of diaphragmatic function with pulmonary function test and thoracic tomodensitometry | up to twenty years after inclusion
  Using Spirometry (Vital capacity in supine position)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Benveniste, PU PH, Study Director — Groupe Hospitalier Pitie-Salpetriere; Yves Allenbach, Study Director — Groupe Hospitalier Pitie-Salpetriere
Locations (2):
- France (2):
  - Département de médecine interne et immunolgie clinique, Hôpital Pitié Salpêtrière, Paris
  - Département de pharmacologie clinique, Hôpital Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Power JR, Dolladille C, Ozbay B, Procureur A, Ederhy S, Palaskas NL, Lehmann LH, Cautela J, Courand PY, Hayek SS, Zhu H, Zaha VG, Cheng RK, Alexandre J, Roubille F, Baldassarre LA, Chen YC, Baik AH, Laufer-Perl M, Tamura Y, Asnani A, Francis S, Gaughan EM, Rainer PP, Bailly G, Flint D, Arangalage D, Cariou E, Florido R, Narezkina A, Liu Y, Sandhu S, Leong D, Issa N, Piriou N, Heinzerling L, Peretto G, Crusz SM, Akhter N, Levenson JE, Turker I, Eslami A, Fenioux C, Moliner P, Obeid M, Chan WT, Ewer SM, Kassaian SE, Johnson DB, Nohria A, Ben Zadok OI, Moslehi JJ, Salem JE; International ICI-Myocarditis Registry. Immune checkpoint inhibitor-associated myocarditis: a novel risk score. Eur Heart J. 2025 Jun 18:ehaf315. doi: 10.1093/eurheartj/ehaf315. Online ahead of print. PMID 40569849
- [Derived] Power JR, Dolladille C, Ozbay B, Procureur AM, Ederhy S, Palaskas NL, Lehmann LH, Cautela J, Courand PY, Hayek SS, Zhu H, Zaha VG, Cheng RK, Alexandre J, Roubille F, Baldassarre LA, Chen YC, Baik AH, Laufer-Perl M, Tamura Y, Asnani A, Francis S, Gaughan EM, Rainer PP, Bailly G, Flint D, Arangalage D, Cariou E, Florido R, Narezkina A, Liu Y, Sandhu S, Leong D, Issa N, Piriou N, Heinzerling L, Peretto G, Crusz SM, Akhter N, Levenson JE, Turker I, Eslami A, Fenioux C, Moliner P, Obeid M, Chan WT, Ewer SM, Kassaian SE; International ICI-Myocarditis Registry; Johnson DB, Nohria A, Zadok OIB, Moslehi JJ, Salem JE. Predictors and Risk Score for Immune Checkpoint-Inhibitor-Associated Myocarditis Severity. medRxiv [Preprint]. 2024 Jun 3:2024.06.02.24308336. doi: 10.1101/2024.06.02.24308336. PMID 38883792